CLINICAL TRIAL: NCT02186626
Title: Phase 1 Study of the Safety and Immunogenicity of a 2-Dose Regimen of West Nile/Dengue 4-3´Δ30 Chimeric Virus Vaccine (WN/DEN4Δ30), a Live Attenuated Vaccine for West Nile Encephalitis, in Flavivirus-naïve Adults 50-65 Years of Age
Brief Title: Evaluating the Safety and Immunogenicity of a Live Attenuated West Nile Virus Vaccine for West Nile Encephalitis in Adults 50 to 65 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 290; WIRB/20140078
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: West Nile Virus
Keywords: West Nile Virus, vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WN/DEN4Δ30 Vaccine (Experimental): Participants will receive one dose of the WN/DEN4Δ30 vaccine at study entry and one dose at Day 180.
  Interventions: Biological: WN/DEN4Δ30 Vaccine
- Placebo (Placebo Comparator): Participants will receive one dose of the placebo at study entry and one dose at Day 180.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: WN/DEN4Δ30 Vaccine — WN/DEN4Δ30 vaccine is a live attenuated, recombinant, chimeric virus. Dose: 10^4 plaque-forming units (PFUs); delivered by subcutaneous injection in the deltoid region of the upper arm.
  Arms: WN/DEN4Δ30 Vaccine
Biological: Placebo — Delivered by subcutaneous injection in the deltoid region of the upper arm.
  Arms: Placebo

SUMMARY:
West Nile virus (WNV) is considered an emerging virus in the United States, and infection can lead to severe illness in older adults. This study will evaluate the safety of and immune response to a live West Nile virus vaccine (WN/DEN4Δ30) for the prevention of West Nile encephalitis in adults 50 to 65 years old.

DETAILED DESCRIPTION:
WNV is the leading vector-borne cause of viral encephalitis in the United States. Severe illness is most common in older adults, and in this population, the virus can cause hepatitis, meningitis, and encephalitis leading to paralysis, coma, and death. WNV illness is a public health issue and is an emerging disease in the United States. This study will evaluate the safety and immunogenicity of a live attenuated West Nile/dengue chimeric virus vaccine (WN/DEN4Δ30) for the prevention of West Nile encephalitis in adults 50 to 65 years old.

This study will enroll healthy adults, 50 to 65 years old, who have no history of previous flavivirus infection. Participants will be randomly assigned to receive the WN/DEN4Δ30 vaccine or placebo vaccine at study entry (Day 0). At the entry visit, participants will undergo a medical history review, physical examination, blood collection, and vital sign measurements; female participants will also take a pregnancy test. Participants will then receive their assigned vaccine, and they will remain in the clinic for 30 minutes after the vaccination for monitoring. Participants will record their temperature and symptoms 3 times a day for 16 days after each vaccination. Additional study visits will occur on Days 3, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, and 150. These visits may include the same study procedures that occurred at the entry visit. At a study visit on Day 180, participants will receive another dose of their assigned vaccine. Additional study visits will occur on Days 183, 186, 188, 190, 192, 194, 196, 201, 208, 236, 270, and 360. All study procedures after the second vaccination will be the same that occurred after the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant, non-breastfeeding females between 50 and 65 years of age, inclusive. Children will not be recruited or enrolled in this study for safety considerations.
* Good general health, as determined by means of the screening procedures
* Available for the duration of the trial
* Willingness to participate in the study as evidenced by signing the informed consent form (ICF)

Exclusion Criteria:

* Pregnancy, as determined by positive beta-human choriogonadotropin (HCG) test (if female)
* Currently lactating and breastfeeding (if female)
* Participant is unwilling to use reliable contraception methods for the duration of the trial (reliable methods of birth control include: pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; surgical sterilization; intrauterine device; abstinence; and post-menopausal documented for at least 1 year). All female participants will be considered as having childbearing potential except for those with documented hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or who are post-menopausal for at least 1 year since last menstrual period.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participant has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* Positive HIV-1 serology by screening and confirmatory assays
* Positive for hepatitis C virus (HCV) by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by positive hepatitis B surface antigen (HBsAg)
* Any confirmed or suspected immunosuppressive or immune modulating disorder (e.g., asplenia, lupus, rheumatoid arthritis, vasculitis, scleroderma, and diabetes mellitus)
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period post-vaccination (topical and nasal steroids are allowed)
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* History of a surgical splenectomy
* Receipt of blood products within the past 3 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* History or serologic evidence of previous WNV infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, and dengue virus)
* Previous receipt of yellow fever, WNV, or dengue vaccine (licensed or investigational)
* Receipt of any investigational agent in the past 28 days or anticipation of receipt of any investigational agent within 28 days following vaccination
* Refusal to allow storage of specimens for future research

Inclusion Criteria for Second Dose:

* Good general health, as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 26 weeks after the second dose
* Ongoing willingness to participate in the study
* Females only: female participants of childbearing potential willing to use effective contraception for the duration of the trial. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than 6 months since last sexual encounter). All female participants will be considered as having childbearing potential except for those with documented hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or who are post-menopausal for least 1 year since last menstrual period.

Exclusion Criteria for Second Dose:

* Anaphylaxis or angioedema following the first dose of vaccine
* Females only: currently pregnant, as determined by positive beta-HCG test, or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* HCV infection, by screening and confirmatory assays
* HBV infection, by HBsAg screening
* Any confirmed or suspected immunosuppressive or immune modulating disorder (e.g., asplenia, lupus, rheumatoid arthritis, vasculitis, scleroderma, or diabetes mellitus)
* Current use of anticoagulant medications
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period post-vaccination (topical and nasal steroids are allowed)
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* History of surgical splenectomy
* Receipt of blood products within the past 3 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* Receipt of any other investigational agent in the 28 days before vaccination or anticipated within 28 days following vaccination
* Refusal to allow storage of specimens for future research

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse events (AEs) | Measured through Day 360
  As classified by both intensity and severity through active and passive surveillance
Measurement of anti-WNV neutralizing antibody | Measured through Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Vaccine Testing Center, University of Vermont College of Medicine (UVM), Burlington, Vermont

REFERENCES:
- [Background] Durbin AP, Wright PF, Cox A, Kagucia W, Elwood D, Henderson S, Wanionek K, Speicher J, Whitehead SS, Pletnev AG. The live attenuated chimeric vaccine rWN/DEN4Delta30 is well-tolerated and immunogenic in healthy flavivirus-naive adult volunteers. Vaccine. 2013 Nov 19;31(48):5772-7. doi: 10.1016/j.vaccine.2013.07.064. Epub 2013 Aug 19. PMID 23968769